CLINICAL TRIAL: NCT02122419
Title: Phase IV Study of Application Position During Spinal Anesthesia
Brief Title: The Effect of Patient Position on Postdural Puncture Headache
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İBRAHİM ÖZTÜRK, doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: PDPHPOSITION
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Pregnancy; Headache
MeSH Terms: conditions — Headache | interventions — Sitting Position

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- lateral: spinal anesthesia performed during lateral position
  Interventions: Other: lateral
- sitting: spinal anesthesia performed during sitting position
  Interventions: Other: sitting

INTERVENTIONS:
Other: lateral — spinal anesthesia performed during lateral position
  Groups: lateral
Other: sitting — spinal anesthesia performed during sitting position
  Groups: sitting

SUMMARY:
We aimed to investigate the association between the position in which spinal anesthesia was performed and postdural puncture headache occurrence.

DETAILED DESCRIPTION:
Records of patients who underwent caesarean section between January, 2013 and November, 2013 with spinal anesthesia will be retrospectively examined. Demographic data of patients, comorbid diseases, position of patient while performing spinal anesthesia, the number of spinal puncture attempts will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years were included

Exclusion Criteria:

* Conversion to general anesthesia was the exclusion criteria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients records form patients who experienced headache after caesarean section with spinal anesthesia were retrospectively evaluated
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
postdural puncture headache | postoperative first day
  patient records will be evaluated regarding post dural puncture headache

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim öztürk, M.D, Principal Investigator — Ministery of Health
Locations (1):
- Dışkapı Yıldırım Beyazıt Education and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Dogan M, Turker H, Ugurlu M, Ergun F, Bozkurt M. Do peroperative supine and prone positions have an effect on postspinal headache incidence? Neurosciences (Riyadh). 2005 Jan;10(1):64-7. PMID 22473188
- [Background] Gil NS, Lee JH, Yoon SZ, Jeon Y, Lim YJ, Bahk JH. Comparison of thoracic epidural pressure in the sitting and lateral decubitus positions. Anesthesiology. 2008 Jul;109(1):67-71. doi: 10.1097/ALN.0b013e31817b80df. PMID 18580174
- [Background] Abel AS, Brace JR, McKinney AM, Friedman DI, Smith SD, Westesson PL, Nascene D, Ott F, Lee MS. Effect of patient positioning on cerebrospinal fluid opening pressure. J Neuroophthalmol. 2014 Sep;34(3):218-22. doi: 10.1097/WNO.0000000000000074. PMID 24213568